CLINICAL TRIAL: NCT04731909
Title: Clinical Study of Toripalimab Combined With Anlotinib, Etoposide and Platinum in the Treatment of Extensive-stage Small Cell Lung Cancer
Brief Title: Toripalimab Combined With Anlotinib, Etoposide and Platinum in the Treatment of Extensive-stage Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, Head of Oncology, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT-SCLC-02
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: SCLC, Extensive Stage; Lung Cancer; Small Cell Lung Cancer
Keywords: Anti-PD-1; Anti-angiogenesis; chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — toripalimab; anlotinib; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With Anlotinib, Etoposide and Platinum (Experimental): Toripalimab 240mg,d1,q3w+Anlotinib 12mg/d,d1-14,q3w+Etoposide 100mg/m2,d1-3,q3w+Cisplatin 75mg/m2 or Carboplatin AUC=5, d1, q3w,4-6 cycles in total. After the end of the first-line treatment, patients with CR, PR, and SD can continue to maintenance treatment with Toripalimab 240mg,d1,q3w+Anlotinib 12mg/d, was taken orally for 2 weeks and stopped for 1 week until the disease progressed.
  Interventions: Drug: Toripalimab; Drug: Anlotinib; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg,ivgtt,d1,q3w.
  Other Names: Toripalimab Injection; Teruipuli dankang Zhusheye; TuoYI; JS001
Drug: Anlotinib — Anlotinib 12 mg/d,d1-14,q3w,4-6 cycles in total. In maintenance treatment period, Anlotinib 12 mg/d,d1,Oral for 2 weeks and stop for 1 week.
  Other Names: Anlotinib Hydrochloride Capsules; FuKeWei
Drug: Cisplatin — 75mg/m2,d1,q3w,4-6 cycles in total.
  Other Names: Cisplatin injection
Drug: Carboplatin — AUC=5,d1,q3w,4-6 cycles in total.
  Other Names: Carboplatin injection

SUMMARY:
To evaluates the effectiveness and safety of Toripalimab combined with Anlotinib and chemotherapy for the first-line treatment of ES-SCLC, and maintenance therapy are Toripalimab combined with Anlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and voluntarily sign informed consent;
2. Age: 18-75 years old;
3. Expected survival period ≥ 3 months;
4. Small cell lung cancer confirmed by histology or cytology, extensive stage disease (American Joint Committee on Cancer (7th edition) stage IV SCLC [any T stage, any N stage and Mla/b]), or T3-4 adult patients(≥18 years old) who cannot be included in a tolerable radiotherapy plan due to a wide range of multiple lung nodules or the tumor/nodule size is too large;
5. According to the RECIST 1.1 standard, the patient has at least one target lesion with a measurable diameter(The long diameter of CT scan of tumor lesions is ≥10 mm, the short diameter of CT scan of lymph node lesions is ≥15 mm, and the scan thickness is not more than 5 mm);
6. ECOG PS: 0-2;
7. Patients with brain metastases must be asymptomatic or stable on treatment with steroids and anticonvulsants within 1 month before study treatment;
8. The patient must be considered suitable for platinum-based chemotherapy as the first-line treatment for SCLC, Chemotherapy must include either cisplatin or carboplatin, combined with etoposide;
9. Laboratory test indicators must meet the following requirements: Hematology: white blood cells ≥4.0×10^9/L, neutrophils ≥2.0×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90g/L. Liver function: serum bilirubin is lower than 1.5 times the maximum normal value; for patients without liver metastasis: ALT and AST are lower than 2.5 times the maximum normal value; for patients with liver metastasis: ALT and AST are lower than 5 times the maximum normal value ; Measured or calculated creatinine clearance: According to the Cockcroft-Gault formula (using actual body weight), patients receiving cisplatin treatment>60mL/min, and patients receiving carboplatin treatment>45mL/min;
10. Good compliance and follow-up;
11. The urine or serum pregnancy test results of premenopausal women were negative.

Exclusion Criteria:

1. Participated in another clinical study within the last 4 weeks and received etoposide + platinum (cisplatin or carboplatin) administration;
2. There is a medical contraindication to etoposide-platinum (carboplatin or cisplatin)-based chemotherapy;
3. Patients who have previously received vascular endostatin (such as bevacizumab, Regorafenib, etc.) ;
4. Allow radiation therapy outside the chest (ie, bone metastases) for the purpose of palliative care;
5. Etoposide + platinum (cisplatin or carboplatin) received major surgery within 28 days before the first dose (defined by the investigator). Note: For the purpose of palliative care, local surgery on isolated lesions is acceptable;
6. Patients with symptomatic brain metastases;
7. People with hypertension who cannot be well controlled by a single antihypertensive drug (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
8. Urine routine test showed urine protein ≥++ and confirmed 24-hour urine protein quantification>1.0g;
9. Cardiovascular disease history: congestive heart failure> New York Heart Association (NYHA) standard II, patients with active coronary artery disease (those with myocardial infarction 6 months before enrollment can be enrolled), arrhythmia requiring treatment (Allows to take beta blockers or digoxin);
10. Active severe clinical infections (>NCI-CTCAE 3.0 version 2 infection criteria), including tuberculosis (clinical evaluation, including clinical history, physical examination, imaging findings and TB examination in line with local clinical practice), hepatitis B (known HBV Surface antigen [HbsAg] positive), hepatitis C or human immunodeficiency virus (HIV 1/2 antibody positive). Patients who have previously had HBV infection or have been cured (defined as the presence of hepatitis B core IgG antibodies and the absence of HBsAg) are eligible. Hepatitis C virus (HCV) antibody-positive patients are only eligible if the HCV RNA polymerase chain reaction is negative;
11. History of allogeneic organ transplantation;
12. Patients with bleeding tendency or coagulation disorders, (14 days before randomization must meet: INR is within the normal range without the use of anticoagulants);
13. In the past 2 years, there are active autoimmune diseases that require systemic treatment (such as corticosteroids or immunosuppressive drugs), and related alternative treatments (such as thyroxine, insulin, or physiological corticosteroid replacement for renal or pituitary insufficiency) are allowed treatment);
14. Those who have received live vaccination within 4 weeks before the start of treatment;
15. Patients requiring renal dialysis;
16. Those who had suffered from tumors other than small cell lung cancer within 5 years before being enrolled in this study. Except: cervical carcinoma in situ, cured basal cell carcinoma, cured bladder epithelial tumor;
17. Arteriovenous thrombosis events occurred within one year before screening, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism, etc.;
18. Pulmonary hemorrhage ≥ CTCAE grade 2 occurred within 4 weeks before the first use of the study drug;
19. Bleeding from other parts of CTCAE Grade 3 or higher within 4 weeks before the first use of the study drug, including the following conditions: local active ulcer lesions and fecal occult blood (+ +); patients with a history of melena and hematemesis within 2 months; researcher People who think that massive gastrointestinal bleeding may occur;
20. Severe unhealed wounds, ulcers or fractures;
21. Uncorrected dehydration;
22. Patients who are pregnant or breastfeeding;
23. Drug abuse and medical, psychological or social conditions may interfere with patient participation in research or have an impact on the evaluation of research results;
24. Known or suspected allergy to the test drug or any drug related to the test given;
25. Any unstable conditions may endanger the safety of patients and affect their compliance with research;
26. Patients with poor compliance;
27. Researchers think it is inappropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to 2 years
  Defined as the time interval from randomization to death. If the patient continues to survive or his life or death is unknown, the date of death will be reviewed using the latest point in time when the patient is still alive.

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 2 years
  It is defined as the number of cases achieving CR, or PR, as a percentage of patients with evaluable efficacy. Disease remission and progress will be evaluated based on RECIST standards.
Disease control rate(DCR) | up to 2 years
  The percentage of cases that achieved remission (PR+CR) and stable disease (SD) after treatment accounted for the number of evaluable cases. In short, DCR=CR+PR+SD. And the RECIST standard is to maintain at least 4 weeks.
Progress Free Survival(PFS) | up to 2 years
  It is defined as the time interval from randomization of patients to disease progression or death, whichever comes first. There was no progress or the time of disease progression was not recorded when the trial was withdrawn, and the date of the last examination was used as the end date.

OTHER OUTCOMES:
Adverse Event (AE) | up to 2 years
  Any untoward medical occurrence that may present during treatment with a pharmaceutical product but which does not necessarily have a causal relationship with this treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, PH.D, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No